CLINICAL TRIAL: NCT06417957
Title: The Effect of Cultural Competence Education Given According to the Peer Education Model on the Cultural Competence Levels of Student Nurses
Brief Title: Cultural Competence Education Given According to the Peer Education Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Cennet Ciriş Yıldız, Asistant Prof., Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1919B012203801
Record Dates: First submitted 2023-01-30; First posted 2024-05-16 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Culture Shock; Cultural Competence
Keywords: cultural knowledge, cultural practice, cultural sensitivity, cultural competence

STUDY DESIGN:
Intervention Model Description: Group 1: Experimental group (Education group) Goup 2: Control group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental group (Education group)
  Interventions: Other: cultural competence training
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: cultural competence training — The peer students in the experimental group will be given a total of 16 hours of cultural competence training, two days a week, two lessons per day (60 min. + 60 min.) for four weeks.
  Arms: Experimental

SUMMARY:
The aim of the study is to determine the effect of cultural competence education given according to the peer education model on the cultural competence levels of student nurses.

DETAILED DESCRIPTION:
Nursing students will be given cultural competence training (with peer education model) and then the effectiveness of this training will be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Not receiving training on cultural competence,
* Participated in Cultural Competence Peer Training for the experimental group,
* Filled out the survey 3 times on the specified dates for the experimental and control groups,
* Volunteer to participate in the research,
* 3rd and 4th year nursing students.

Exclusion criteria:

* Receiving training on cultural competence,
* Not participating in Cultural Competency Peer Training for the experimental group,
* Failure to fill out the survey 3 times on the specified dates for the experimental and control groups,
* Those who do not volunteer to participate in the research,
* 1st and 2nd year nursing students,
* Students who want to leave the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Cultural Competence Assessment Tool | Before training, immediately in the first and third months after training
  Cultural Qualıfıcatıon Assessment Scale (Special For Nursing Students). The level of cultural competence is determined by scoring the scale for four dimensions (cultural awareness, cultural knowledge, cultural sensitivity, cultural practice) with a specific score chart. cultural competence In determining the level, if one of the KYDS items is marked as "strongly agree" or "agree", the answer is considered correct and one (1) point is received; If "disagree" or "strongly disagree" is marked, the answer is considered incorrect and zero (0) points are received and the points are added up. The score that can be obtained from each dimension varies between 0-10. The maximum score that can be obtained from the total score of the four dimensions of the scale is forty (40). Scoring 40 points from the scale indicates that the individual is "culturally competent".

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No